CLINICAL TRIAL: NCT01077739
Title: A Single-arm Open-label Phase II Study: Treatment Beyond Progression by Adding Bevacizumab to XELOX or FOLFOX Chemotherapy in Patients With Metastatic Colorectal Cancer and Disease Progression Under First-line FOLFIRI + Bevacizumab Combination
Brief Title: A Study of Avastin (Bevacizumab) With XELOX or FOLFOX in Patients With Metastatic Colorectal Cancer and Disease Progression Under First-line FOLFIRI and Avastin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22519; 2009-012090-36; NCT01069679 (obsolete NCT alias)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Bevacizumab; Capecitabine; Oxaliplatin

ARMS (1):
- Avastin (bevacizumab) + standard of care (Experimental)
  Interventions: Drug: fluorouracil (5FU); Drug: leucovorin; Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: oxaliplatin

INTERVENTIONS:
Drug: fluorouracil (5FU) — standard FOLFOX regimen
Drug: leucovorin — standard FOLFOX regimen
Drug: bevacizumab [Avastin] — 7.5 mg/kg iv infusion every 3 weeks OR 5 mg/kg iv infusion every 2 weeks
Drug: capecitabine [Xeloda] — standard XELOX regimen
Drug: oxaliplatin — standard XELOX or FOLFOX regimen

SUMMARY:
This open-label single arm study will evaluate the efficacy and safety of Avastin added to XELOX or FOLFOX in patients with metastatic colorectal cancer and disease progression on 1st line therapy with FOLFIRI plus Avastin. Patients will receive either Avastin (7.5mg/kg iv infusion every 3 weeks) and standard XELOX (Xeloda [capecitabine] plus oxaliplatin) chemotherapy or Avastin (5 mg/kg iv infusion every 2 weeks) and standard FOLFOX (5-FU and leucovorin plus oxaliplatin) chemotherapy. The anticipated time on study treatment is until disease progression, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/=18 years of age
* metastatic colorectal cancer
* at least 1 measurable lesion according to RECIST v. 1.1
* patients with disease progression with prior FOLFIRI + Avastin therapy who are not candidates for primary metastasectomy
* disease progression </= 8 weeks after last dose of Avastin
* ECOG </=2
* No more than 8 weeks between 1st-line treatment with FOLFIRI + Avastin and 2nd-line treatment with XELOX or FOLFOX + Avastin

Exclusion Criteria:

* disease progression > 8 weeks after last Avastin administration
* clinically significant cardiovascular disease
* CNS disease except for treated brain metastasis
* history of other malignancies within 2 years prior to start of study treatment (with the exception of curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix)
* major surgery, open biopsy, or significant traumatic injury within 28 days prior to start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Belgium (26):
  - Aalst
  - Arlon
  - Assebroek
  - Aye
  - Bonheiden
  - Brasschaat
  - Bruges
  - Brussels
  - Charleroi
  - Dendermonde
  - Edegem
  - Genk
  - Ghent
  - Hasselt
  - Kortrijk
  - Mechelen
  - Merksem
  - Mont-godinne
  - Montigny-le-Tilleul
  - Namur
  - Ostend
  - Sint-Niklaas
  - Tournai
  - Turnhout
  - Verviers
  - Wilrijk

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Oxaliplatin + Capecitabine: Participants received bevacizumab 7.5 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1; oxaliplatin 130 mg per square meter (mg/m^2) IV on Day 1; and capecitabine 1000 mg/m^2, orally (PO), twice daily (BID) on Days 1 through 14 (followed by 1-week rest period). The cycle was repeated every 3 weeks until disease progression.
- Bevacizumab + 5-fluorouracil/Oxaliplatin/Leucovorin (FOLFOX): Participants received bevacizumab 5.0 mg/kg IV on Day 1 and FOLFOX (5-fluorouracil [5-FU] plus leucovorin and oxaliplatin) administered on Days 1 and 2 (followed by a rest period on Days 3 through 14); the specific FOLFOX regimen was determined on an individual participant basis by the investigator (5-FU and leucovorin dose was dependent on choice of FOLFOX regimen; oxaliplatin was administered at a dose ranging from 85 to 130 mg/m^2 IV on Day 1 based on choice of FOLFOX regimen). The cycle was repeated every 2 weeks until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + 5-fluorouracil/Oxaliplatin/Leucovorin (FOLFOX)
Started | 25 | 50
Completed | 20 | 40
Not Completed | 5 | 10
Not completed — Premature withdrawal | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 3
Not completed — Unacceptable toxicity | 1 | 2
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all enrolled participants who received at least 1 dose of the investigational and non-investigational products.
Groups:
- Bevacizumab + Oxaliplatin + Capecitabine: Participants received bevacizumab 7.5 mg/kg IV on Day 1; oxaliplatin 130 mg/m^2 IV on Day 1; and capecitabine 1000 mg/m^2, PO, BID on Days 1 through 14 (followed by 1-week rest period). The cycle was repeated every 3 weeks until disease progression.
- Bevacizumab + FOLFOX: Participants received bevacizumab 5.0 mg/kg IV on Day 1 and FOLFOX (5-FU plus leucovorin and oxaliplatin) administered on Days 1 and 2 (followed by a rest period on Days 3 through 14); the specific FOLFOX regimen was determined on an individual participant basis by the investigator (5-FU and leucovorin dose was dependent on choice of FOLFOX regimen; oxaliplatin was administered at a dose ranging from 85 to 130 mg/m^2 IV on Day 1 based on choice of FOLFOX regimen). The cycle was repeated every 2 weeks until disease progression.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX | Total
Number analyzed (Participants) | 25 | 50 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.9) | 64.9 (8.7) | 63.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 21 | 29
  Male | 17 | 29 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) From the Start of Treatment Beyond Progression
Description: PFS from the start of treatment beyond progression was defined as the interval between the start of beyond-progression therapy and the date at which disease progression was documented. Progression of disease was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 and abdominal/pelvic computerized tomography (CT) or magnetic resonance imaging (MRI) scanning as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The same method of assessment and the same technique were to be used to evaluate each lesion throughout the entire study. If more than one method was used, data from the most accurate method according to RECIST were recorded. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks until disease progression, at end of treatment or withdrawal, for up to 24 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX
Number analyzed (Participants) | 25 | 50
months | 6.3 [4.1 to 7.6] | 5.1 [3.8 to 6.0]

2. Secondary Outcome: PFS From the Start of First-Line Therapy
Description: PFS from the start of first-line therapy was defined as the interval between the start of first-line therapy and the date at which second disease progression (after the start of beyond progression therapy) was documented. Progression of disease was evaluated using RECIST version 1.1 and abdominal/pelvic CT or MRI scanning. The same method of assessment and the same technique were to be used to evaluate each lesion throughout the entire study. If more than one method was used, data from the most accurate method according to RECIST were recorded. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks until disease progression, at end of treatment or withdrawal, for up to 24 months
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX
Number analyzed (Participants) | 25 | 50
months | 17.8 [14.1 to 19.4] | 18.0 [15.0 to 19.9]

3. Secondary Outcome: Percentage of Participants With an Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Percentage of participants with an overall response of CR or PR according to RECIST criteria.
  CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<]10 millimeters [mm]). No new lesions. PR was defined as greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 9 weeks until disease progression, at end of treatment or withdrawal, for up to 24 months
Population: ITT population; only participants with RECIST evaluations were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX
Number analyzed (Participants) | 22 | 47
percentage of participants | 27.3 | 6.4

4. Secondary Outcome: Geometric Mean Values of Pro-Angiogenic Cytokine Concentrations at Baseline and Prior to Progression
Description: Pro-angiogenic cytokine concentrations of placental growth factor (PlGF), basic fibroblast growth factor (bFGF), and hepatocyte growth factor (HGF) in participant sera were measured and reported in units of picograms/milliliter (pg/mL). The geometric mean was calculated as exp10 (mean of log10 transformed concentration) and the standard deviation (SD) is SD of log10 transformed concentration.
Time Frame: Baseline, every 9 weeks until disease progression, at final visit or at withdrawal, for up to 24 months
Population: ITT Population. Number (n) equals (=) number of participants assessed for the given parameter at the specified visit.
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX
Number analyzed (Participants) | 13 | 23
pg/mL
  Baseline bFGF (n=13,23) | 6.8 (0.7) | 6.1 (0.6)
  bFGF, Prior to progression levels (n=12,18) | 3.6 (0.9) | 4.2 (0.7)
  Baseline HGF (n=13,23) | 133.0 (0.3) | 186.0 (0.4)
  HGF, Prior to progression levels (n=12,18) | 187.3 (0.4) | 230.3 (0.4)
  Baseline PIGF (n=13,23) | 29.8 (0.1) | 26.3 (0.2)
  PIGF, Prior to progression levels (n=12,18) | 34.7 (0.1) | 37.1 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from Day 1 until 28 days after last dose of study medication for up to 24 months.
Description: The safety population included all participants who received at least 1 dose of the investigational or non-investigational products.
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine | Bevacizumab + FOLFOX
Serious Adverse Events (participants affected / at risk) | 12/25 | 18/50
Other Adverse Events (participants affected / at risk) | 24/25 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Oxaliplatin + Capecitabine (N=25) | Bevacizumab + FOLFOX (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 3
Idiosyncratic drug reaction (General disorders) | 0 | 1
Obstruction (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Vaginal abscess (Infections and infestations) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Oxaliplatin + Capecitabine (N=25) | Bevacizumab + FOLFOX (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 8
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 7
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 13
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 14 | 21
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 16
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 2
Rectal tenesmus (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Steatorrhoea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5
Asthenia (General disorders) | 5 | 7
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 9 | 22
Feeling cold (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 1 | 2
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 2 | 4
Pyrexia (General disorders) | 3 | 8
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 5
Hypersensitivity (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 1 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 1
Tracheitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Weight decreased (Investigations) | 3 | 2
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 2 | 2
Memory impairment (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 7 | 9
Neurotoxicity (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 6 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0
Polyneuropathy (Nervous system disorders) | 3 | 7
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Apathy (Psychiatric disorders) | 0 | 2
Disorientation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2
Renal pain (Renal and urinary disorders) | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 13
Vascular insufficiency (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.